CLINICAL TRIAL: NCT03565198
Title: Serum Ferritin as a Predictor for Development of Anemia in Pregnancy: A Pilot Study
Brief Title: Ferritin as a Predictor for Anemia in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Paul Dietz, PI, CAMC Health System
Other Study IDs: 17-366
Record Dates: First submitted 2018-06-12; First posted 2018-06-21 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Anemia, Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2.5 mL aliquots of serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anemia is a common problem with pregnant women around the world. There are high rates even within industrialized nations. The main cause of anemia in pregnancy is a lack of iron. There have been medical programs that give iron vitamins to all pregnant patients at the beginning of care to decrease anemia. These programs did not adequately decrease anemia in pregnancy. Many of them gave iron vitamins in doses that were low because pregnant patients sometimes have side effects to it. The next idea was to figure out which women were more at risk to get anemia and then treat them with a higher amount of iron. There are different blood tests to see how much iron stores are in the blood, but many do not work well during pregnancy. The test study staff think is the best for this is ferritin. The goal of this first small study is to see if healthcare providers can use the level of ferritin to predict anemia in pregnancy. This would then help to better screen, diagnose, and treat anemia during pregnancy. Study staff will enroll obstetric patients from the Women's Medicine Center and compare ferritin levels in these patients early in pregnancy with diagnosis of anemia later in pregnancy.

DETAILED DESCRIPTION:
In the past, all pregnant patients were started on an iron supplement (in addition to that which is in prenatal vitamins), with the presumption that they had low or inadequate iron stores. That "habit" has gone by the wayside. Now, health care providers wait until a patient is already anemic and then start iron supplementation. In general, the first opportunity to determine if a patient is anemic as the pregnancy progresses comes at about 28 weeks of gestation when routine laboratory testing includes a Hemoglobin level. It is the author's hope that there is some middle ground.

d. Specific Aims/Objectives:

The aim of this study is to test if ferritin levels taken in early pregnancy can predict the development of iron deficiency anemia later in pregnancy.

Hypothesis: Serum ferritin levels, when tested prior to 20 weeks gestation, can identify women who will develop iron deficiency anemia before delivery.

e. Methods, Procedure, Sample

Design: This is a prospective pilot study to test for anemia in a cohort of pregnant women.

Sample:

Participants will be recruited for participation from the Women's Medicine Center at Charleston Area Medical Center's Women and Children's Hospital in Charleston, WV. Enrollment will continue until a sufficient sample size is attained. A total of 130 obstetric patients will be enrolled in this pilot study with the target of a final sample size of 100 (lab work completed). Based on an anemia prevalence of 35% at this institution and accounting for a potential loss to follow up rate around 23%, study staff expect to have 35 women test positive for anemia (defined as Hgb < 11 g/dL). There is no published data in the literature regarding ferritin in the first trimester to predict anemia.

The following inclusion/exclusion criteria will be applied:

Inclusion criteria:

* Age 15-45 years old at intake
* Confirmed intrauterine pregnancy by 1st trimester ultrasound

Exclusion criteria:

* Antepartum iron supplementation, other than prenatal vitamins
* Placental abruption or hemorrhage
* Initial visit >20 weeks gestation
* Diagnosis of sickle cell disease or thalassemia
* Diagnosed with anemia at initial prenatal visit
* Diagnosis of autoimmune issues that could effect iron levels

Data Collection/Instrumentation

Patients will be enrolled in this study through the resident and midwife clinics at the Women's Medicine Center. Staff from the Charleston Area Medical Center Health Education and Research Institute Outcomes Research will obtain consent from interested obstetric patients. All patients in this clinic undergo routine laboratory testing that comprises a standard "Prenatal Panel" following their intake prenatal visit. This includes universal screening for anemia. Willing participants will have a serum ferritin level added to this laboratory panel, which will not result in any deviation from standard care or additional phlebotomy. An amount of 2.5 mL aliquots of serum per study participant will be used for study analysis and will be stored in a -30 degree Centigrade freezer until a sample size of 130 participants is met. All samples will then be processed simultaneously, which will likely reduce inter-assay variability. 2µL of serum will be processed using SIEMENS Dimension Vista® System. The results will be expressed as the concentration of ferritin in ng/mL[µg/L] (9). Participants will not be charged any additional fee for having the serum ferritin level added to their laboratory panel.

Patients in the study will continue with routine prenatal care and testing, which includes a repeat Complete Blood Count around 28 weeks gestation. The study will conclude once the final participant completes her 28 week standard lab draw. The hospital and clinic records of all participants will be reviewed once all patients in the study have delivered. Any documentation of significant antepartum blood loss, such as placental abruption or trauma, will exclude patients from the data analysis unless clinical anemia was documented prior to the event. All hemoglobin values obtained during the antepartum period will be used in the final data analysis. These values will come from standard outpatient laboratory testing ordered by healthcare providers, as well as any visits to the antepartum triage unit or hospital admissions. Clinical anemia will be defined based upon the World Health Organization definition of a hemoglobin level that is less than 11 mg/dL. The data will be used to determine if patients who have a low serum ferritin will go on to develop anemia at some point during their antenatal course.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-45 years old at intake
* Confirmed intrauterine pregnancy by 1st trimester ultrasound

Exclusion Criteria:

* Antepartum iron supplementation, other than prenatal vitamins
* Placental abruption or hemorrhage
* Initial visit >20 weeks gestation
* Diagnosis of sickle cell disease or thalassemia
* Diagnosed with anemia at initial prenatal visit
* Diagnosis of autoimmune issues that could effect iron levels

Ages: 15 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Participants will be enrolled through hospital's obstetric clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
clinical anemia | 28 weeks gestation
  hemoglobin < 11 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dietz, MD, Principal Investigator — CAMC
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD data